CLINICAL TRIAL: NCT01077700
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Study of the Safety and Efficacy of ABT-288 in the Treatment of Cognitive Deficits in Schizophrenia (CDS)
Brief Title: Efficacy and Safety Study for Cognitive Deficits in Adult Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-503
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2013-01

CONDITIONS: Cognitive Deficits in Schizophrenia
MeSH Terms: interventions — 2-(4'-(5-methylhexahydropyrrolo(3,4-b)pyrrol-1-yl)biphenyl-4-yl)-2H-pyridazin-3-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-288 Dose 1 (Experimental): low dose of ABT-288
  Interventions: Drug: ABT-288 Low Dose
- ABT-288 Dose 2 (Experimental): high dose of ABT-288
  Interventions: Drug: ABT-288 High Dose
- Sugar Pill (Placebo Comparator): inactive substance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-288 Low Dose
  Arms: ABT-288 Dose 1
Drug: Placebo — inactive substance
  Arms: Sugar Pill
Drug: ABT-288 High Dose
  Arms: ABT-288 Dose 2

SUMMARY:
This is an efficacy and safety study evaluating an experimental treatment for cognitive deficits in adults with schizophrenia.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the efficacy and safety of ABT-288 in approximately 210 adults with schizophrenia. Subjects will be randomized to one of three treatment groups (ABT-288 Dose 1, ABT-288 Dose 2 or placebo) for a 12-week Treatment Period. The purpose of this research study is to find out whether ABT-288 compared to placebo can improve cognition and what side effects ABT 288 may cause. Cognition is the way a person thinks, and it includes abilities like paying attention, focusing, remembering things, and solving problems. Acronyms listed in the Outcomes and/or Eligibility sections for this study are defined below:

* MCCB: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery
* UPSA-2: University of California at San Diego (UCSD) Performance-Based Skills Assessment-2
* CANTAB: Cambridge Neuropsychological Test Automated Battery
* PANSS: Positive and Negative Syndrome Scale
* NSA-16: Negative Symptom Assessment-16
* CGI-S: Clinical Global Impression - Severity

ELIGIBILITY:
Inclusion Criteria:

* Has current DSM-IV-TR diagnosis of schizophrenia confirmed by the Mini-International Neuropsychiatric Interview.
* Is clinically stable while receiving antipsychotic therapy with one or two atypical antipsychotic medications: lack of hospitalizations from 4 months of Initial Screening Visit; taking same antipsychotic medication(s) for at least 8 weeks prior to the Day -1 visit; core positive symptoms of PANSS no worse than moderate in severity throughout Screening Period of at least 4 weeks.
* Has been diagnosed with or treated for schizophrenia for at least 2 years prior to Initial Screening Visit.
* Has had continuity in psychiatric care (e.g., mental health system, clinic or physician) for at least 6 months prior to Initial Screening Visit.
* Has an identified responsible contact person (e.g., family member, social worker, case worker, or nurse) that can provide support to the subject and ensure compliance with protocol requirements.

Exclusion Criteria:

* Has valid current or past diagnosis of schizoaffective disorder, bipolar disorder, manic episode, dementia, posttraumatic stress disorder, obsessive compulsive disorder, or a current major depressive episode.
* Has history of substance abuse (excluding nicotine or tobacco products) or alcohol abuse within 6 months prior to Screening Visit; has a substance dependence disorder (excluding nicotine or tobacco products) that has not been remitted for at least 1 year prior to Initial Screening Visit.
* Is taking any medication for extrapyramidal symptoms at any time from the Initial Screening Visit until the Day -1 Visit.
* Is taking any antidepressant that is excluded, including tricyclic antidepressants and monoamine oxidase inhibitors, at any time from 8 weeks prior to the Day -1 Visit.
* Has significant suicidal ideation at Initial Screening Visit.
* Has had a suicide attempt within 1 year prior to the Day -1 Visit.
* Has participated in another trial utilizing the MATRICS Consensus Cognitive Battery (MCCB) or UCSD Performance-Based Skills Assessment (UPSA) (any version) within 6 months prior to Initial Screening Visit.
* Is currently enrolled in any form of cognitive remediation training.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Cognition: MCCB | Measurements from screening period through 12-week treatment period

SECONDARY OUTCOMES:
Functioning: UPSA-2 | Measurements from screening period through 12-week treatment period
Cognition: CANTAB | Measurements from screening period through 12-week treatment period
Symptom Severity: PANSS, NSA-16, CGI-S | Measurements from screening period through 12-week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: George Haig, PharmD, Study Director — AbbVie
Locations (24):
- United States (24):
  - Site Reference ID/Investigator# 21662, Anaheim, California
  - Site Reference ID/Investigator# 21683, Garden Grove, California
  - Site Reference ID/Investigator# 21581, National City, California
  - Site Reference ID/Investigator# 45310, Norwalk, California
  - Site Reference ID/Investigator# 26400, Pasadena, California
  - Site Reference ID/Investigator# 21584, Pico Rivera, California
  - Site Reference ID/Investigator# 45312, Riverside, California
  - Site Reference ID/Investigator# 45309, San Diego, California
  - Site Reference ID/Investigator# 46603, Plantation, Florida
  - Site Reference ID/Investigator# 21681, Chicago, Illinois
  - Site Reference ID/Investigator# 26397, Shreveport, Louisiana
  - Site Reference ID/Investigator# 21761, Pittsfield, Massachusetts
  - Site Reference ID/Investigator# 21591, St Louis, Missouri
  - Site Reference ID/Investigator# 26409, Brooklyn, New York
  - Site Reference ID/Investigator# 21588, Cedarhurst, New York
  - Site Reference ID/Investigator# 21589, Dayton, Ohio
  - Site Reference ID/Investigator# 26407, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 21601, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 26399, Charleston, South Carolina
  - Site Reference ID/Investigator# 21590, Austin, Texas
  - Site Reference ID/Investigator# 21582, Austin, Texas
  - Site Reference ID/Investigator# 26406, DeSoto, Texas
  - Site Reference ID/Investigator# 26402, Houston, Texas
  - Site Reference ID/Investigator# 27502, Bellevue, Washington

REFERENCES:
- [Result] Haig GM, Bain E, Robieson W, Othman AA, Baker J, Lenz RA. A randomized trial of the efficacy and safety of the H3 antagonist ABT-288 in cognitive impairment associated with schizophrenia. Schizophr Bull. 2014 Nov;40(6):1433-42. doi: 10.1093/schbul/sbt240. Epub 2014 Feb 10. PMID 24516190
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500